CLINICAL TRIAL: NCT02640820
Title: A Prospective, Phase 2a Study to Evaluate the Effectiveness and Safety of DPCP Ointment (Samcyprone™) on the Clearance of Verruca Vulgaris (Common Warts) in Subjects Ages 18 - 65 Years
Brief Title: Evaluate the Effectiveness and Safety of DPCP Ointment (Samcyprone™) on the Clearance of Verruca Vulgaris (Common Warts)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RXi Pharmaceuticals, Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RXI-SCP-1502
Record Dates: First submitted 2015-12-18; First posted 2015-12-29 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Common Warts; HPV (Human Papillomavirus); Periungual Warts; Plantar Warts
Keywords: HPV; Verruca Vulgaris
MeSH Terms: conditions — Warts; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sensitization Phase (Experimental): Up to two doses of Sensitizing DPCP Ointment will be applied and subjects who exhibit a sensitization response will enter the Treatment Phase. Pharmacokinetics (PK) of Sensitizing DPCP Ointment will be measured in a subset of subjects. For PK, blood will be collected prior to application of the Sensitizing DPCP Ointment and again at 1, 2, and 24 hours after application.
  Interventions: Drug: Sensitizing DPCP Ointment
- Treatment Phase (Experimental): In the Treatment Phase, subjects will receive doses of Treatment DPCP Ointment weekly for 10 weeks. Subjects who at the end of the Treatment Phase have exhibited partial clearance of warts may be given the option to continue with an additional 10 weekly treatments.
  Interventions: Drug: Treatment DPCP Ointment

INTERVENTIONS:
Drug: Sensitizing DPCP Ointment — Sensitization
  Other Names: Samcyprone™
  Arms: Sensitization Phase
Drug: Treatment DPCP Ointment — Treatment
  Other Names: Samcyprone™
  Arms: Treatment Phase

SUMMARY:
Warts are benign epidermal tumors caused by human papillomaviruses (HPVs). The active pharmaceutical ingredient DPCP has been used for many years as a compounded formulation in acetone for the treatment of warts, alopecia areata and more recently, cutaneous metastatic melanoma lesions. An improved topical ointment formulation of DPCP called Samcyprone™ will be evaluated for the treatment of common warts.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18 and 65 years of age, inclusive
* Subjects presenting with at least one verruca vulgaris (common cutaneous, plantar, and periungual) warts for at least 4 weeks, but no more than 3 years
* Subject's common warts for treatment must measure between 3 and 20 mm and be located on hands, feet, limbs and/or trunk. A maximum of four (4) cutaneous single warts or one (1) area of clustered or adjacent warts up to 80 mm will be treated

Exclusion Criteria:

* Genital warts may not be selected as target warts
* Subjects that are immuno-compromised
* Presence of systemic or localized diseases, conditions, or medications that could interfere with assessment of safety and efficacy or that compromise immune function

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-12; Primary Completion 2018-01 (Actual); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of Sensitizing DPCP Ointment in eliciting a sensitization response in healthy subjects with common warts by assessing the immunotherapeutic response | 4 to 6 weeks
  Assessment of immunotherapeutic response per subject will include gauging the Delayed-Type Hypersensitivity (DTH) response after application sensitizing DPCP ointment. A minimum +2 DTH response will be considered a positive sensitization result
The effectiveness of Treatment DPCP Ointment will be measured by the Investigator's Global Assessment Score (IGAS) | 11 to 20 weeks
  The Investigator's Global Assessment Score (IGAS) is a 4-point scale that will be used to evaluate wart clearance for all treated warts separately. Results will further be utilized to determine overall clearance of treated warts in total. Wart lesion surface area will be measured and used to assist in determining IGAS Score.

SECONDARY OUTCOMES:
The safety and tolerability of a treatment regimen for common warts consisting of a sensitization dose with Sensitizing DPCP Ointment and ten weekly treatments with Treatment DPCP Ointment, assessed by reported adverse events | 30 weeks
  Reported adverse events and clinically-relevant changes in laboratory testing after treatment will be monitored for severity and frequency; incidence of Treatment-Emergent Adverse Events will be assessed
To evaluate Cmax by pharmacokinetics (PK) of DPCP in blood after topical administration of the Sensitizing DPCP Ointment in a subset of subjects | 2 days
  Determine Cmax of Sensitizing DPCP Ointment in whole blood
To evaluate the time to Cmax by pharmacokinetics (PK) of DPCP in blood after topical administration of the Sensitizing DPCP Ointment in a subset of subjects | 2 days
  Determine the time of Cmax of Sensitizing DPCP Ointment in whole blood
To evaluate the time to last measurable concentration (Tlast) by pharmacokinetics (PK) of DPCP in blood after topical administration of the Sensitizing DPCP Ointment in a subset of subjects | 2 days
  Determine Tlast of Sensitizing DPCP Ointment in whole blood
To evaluate the concentration corresponding to Tlast (Clast) by pharmacokinetics (PK) of DPCP in blood after topical administration of the Sensitizing DPCP Ointment in a subset of subjects | 2 days
  Determine Clast of Sensitizing DPCP Ointment in whole blood
To evaluate the area under the concentration curve (AUC) by pharmacokinetics (PK) of DPCP in blood after topical administration of the Sensitizing DPCP Ointment in a subset of subjects | 2 days
  Determine the AUC of Sensitizing DPCP Ointment in whole blood

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Pavco, PhD, Study Director — RXi Pharmaceuticals
Locations (4):
- United States (4):
  - International Dermatology Research, Miami, Florida
  - Summit Dermatology, Oakbrook Terrace, Illinois
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - Mount Sinai - St. Luke's, New York, New York

IPD SHARING:
Plan to Share IPD: No